CLINICAL TRIAL: NCT03603704
Title: A Single Ascending Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LY3209590 in Japanese Patients With Type 2 Diabetes Mellitus
Brief Title: A Study of LY3209590 in Japanese Participants With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 16552; I8H-JE-BDCF (Other: Eli Lilly and Company)
Record Dates: First submitted 2018-07-18; First posted 2018-07-27 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Cohort 3 is open-label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- LY3209590 (Experimental): Insulin naïve participants with Type 2 Diabetes Mellitus received 5 mg and 10 mg LY3209590 administered subcutaneously (SC) in Cohort 1 and 2 respectively.
  Participants with T2DM received 20 mg LY3209590 administered subcutaneously in Cohort 3.
  Interventions: Drug: LY3209590
- Placebo (Active Comparator): Participants from Cohort 1 and 2 received Placebo administered SC.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3209590 — Administered SC
  Arms: LY3209590
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the safety of a study drug known as LY3209590 in Japanese participants with type 2 diabetes. Side effects and tolerability will be documented. Blood samples will be taken to compare how the body handles the drug and how it affects blood sugar levels. The study will last about four weeks, not including screening. Screening is required within 4 weeks before the start of the study.

ELIGIBILITY:
Inclusion Criteria:

* Have T2DM diagnosed at least 1 year ago
* Have hemoglobin A1c (HbA1c) ≥7.0% and ≤10.0% with fasting plasma glucose (FPG) ≥126 milligrams per deciliter (mg/dL) or HbA1c ≥6.5% and <7.0% with FPG ≥144 mg/dL at screening
* Have body weight ≥54 kilograms and a body mass index >18.5 and ≤40.0 kilograms per square meter at screening

Exclusion Criteria:

* Have received a total daily dose of insulin >1.2 units per kilogram at screening
* Have taken any glucose-lowering medications, other than basal insulin, metformin and dipeptidyl peptidase-IV inhibitor, in the past 3 months before screening
* Have a history of multiple and/or severe allergies to drugs or foods, or a history of severe anaphylactic reaction
* Have a history of heart block or a repeated demonstration of abnormality in the 12-lead electrocardiogram at screening, which in the opinion of the investigator, increases the risks associated with participating in the study

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-08-17 (Actual); Primary Completion 2019-05-27 (Actual); Study Completion 2019-05-27 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline through Day 28
  A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum Observed Concentration (Cmax) of LY3209590 | Baseline through Day 28
  PK: Cmax of LY3209590
PK: Area Under the Concentration Versus Time Curve (AUC) of LY3209590 | Baseline through Day 28
  PK: AUC of LY3209590
Pharmacodynamics (PD): Change from Baseline in Fasting Plasma Glucose | Baseline through Day 15
  PD: Change from Baseline in Fasting Plasma Glucose

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- Japan (3):
  - P-one clinic, Hachiōji, Tokyo
  - Sumida Hospital, Sumida-ku, Tokyo
  - Hakata Clinic, Fukuoka

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nasu R, Oura T, Ohwaki K, Imori M, Furihata K. Pharmacokinetic and Pharmacodynamic Properties of Once-Weekly Insulin Efsitora Alfa in Japanese Patients with Type 2 Diabetes. Diabetes Ther. 2025 Mar;16(3):513-526. doi: 10.1007/s13300-025-01695-x. Epub 2025 Feb 10. PMID 39928225